CLINICAL TRIAL: NCT06673017
Title: A Phase Ib Dose Escalation/Dose Expansion Study of PTM-101 as an Adjunct to Neoadjuvant Therapy for Treatment Naïve, Borderline Resectable and Locally Advanced Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: PTM-101 in Pancreatic Ductal Adenocarcinoma (PDAC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PanTher Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PT-22-001
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Borderline Resectable Pancreatic Adenocarcinoma; Locally Advanced Pancreatic Adenocarcinoma; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a multi-center, non-randomized, single-arm, open-label, phase Ib dose escalation/dose expansion study of PTM-101 in subjects with pancreatic ductal adenocarcinoma (PDAC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Dose escalation will follow a modified (3+3) design to establish the preliminary RP2D and characterize the safety and pharmacokinetic profile of PTM-101, which will be taken together with all prior clinical data to establish and characterize the preliminary RP2D. A maximum of 12 subjects with treatment-naïve, borderline resectable or locally advanced PDAC will be recruited and receive PTM-101 combined with standard of care neoadjuvant chemotherapy, and be followed for a minimum of 24 months.
  Interventions: Drug: PTM-101
- Dose Expansion (Experimental): The dose of PTM-101 will be the preliminary RP2D determined from all available clinical data. Up to 20 subjects, inclusive of those already assigned to the preliminary RP2D in the dose escalation part, with treatment-naïve, borderline resectable or locally advanced PDAC will be recruited and receive PTM-101, combined with standard of care neoadjuvant chemotherapy, and be followed for a minimum of 24 months.
  Interventions: Drug: PTM-101

INTERVENTIONS:
Drug: PTM-101 — PTM-101, an absorbable drug product containing paclitaxel

SUMMARY:
This is a multi-center, non-randomized, single-arm, open-label, phase Ib, dose escalation/dose expansion study of PTM-101 when combined with neoadjuvant chemotherapy for the treatment of treatment-naïve subjects with borderline resectable and locally advanced pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
This is a multi-center, non-randomized, single-arm, open-label, phase Ib dose escalation/dose expansion study of PTM-101 in subjects with pancreatic ductal adenocarcinoma (PDAC). Dose escalation will assess the safety of PTM-101 containing escalating doses of paclitaxel to establish the preliminary Recommended Phase II Dose (RP2D) when combined with neoadjuvant chemotherapy for subjects who are treatment-naïve, have borderline resectable or locally advanced PDAC and are eligible for neoadjuvant chemotherapy. Subsequently, the dose expansion portion will expand the number of subjects at the preliminary RP2D to assess the efficacy of PTM-101.

ELIGIBILITY:
Inclusion Criteria:

* Imaging consistent with primary PDAC (if PDAC is to be confirmed at study-mandated laparoscopy) or imaging consistent with primary PDAC with prior biopsy/cytology
* No radiographic or physical exam evidence of metastatic disease
* No prior chemo-, radio-, or surgical therapy for PDAC
* Acceptable laboratory values
* CA 19-9 <500 U/mL at baseline after biliary decompression
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Ability to provide informed consent
* No signs or symptoms of pancreatitis
* No other active medical issues which would confound interpretation of safety monitoring, efficacy results or prevent the subject from study participation
* Subjects with childbearing potential must agree to use adequate contraception throughout study participation

Exclusion Criteria:

* Active non-pancreatic cancer that currently requires treatment or is being treated; diagnosis of another malignancy within the past 2 years (excluding a history of carcinoma in situ of the cervix, superficial non-melanoma skin cancers, or superficial bladder cancer that has been adequately treated, or stage 1 prostate cancer that does not require treatment or requires only treatment with luteinizing hormone-releasing hormone agonists or antagonists if initiated at least 30 days prior to screening)
* Contraindications or allergies to paclitaxel, PLGA (poly(lactic-co-glycolic ) acid), or contraindications to implantation of PTM-101 or chemotherapies in protocol (e.g., FOLFIRINOX, gemcitabine, nab-paclitaxel)
* Known human immunodeficiency virus (HIV) or active viral hepatitis
* Active ongoing infection or autoimmune disease which may preclude laparoscopy, placement of PTM-101, administration of chemotherapy or surgical resection of pancreatic tumor
* Inability to comply with activities and therapeutic interventions as outlined in the schedule of events
* Currently enrolled in another investigational drug or device trial
* Women who are pregnant or breastfeeding or who plan to become pregnant or breastfeed; men who plan to donate sperm or conceive a child
* Any other medical or surgical conditions, including prior abdominal surgery, that would preclude safe laparoscopy or implantation in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation | Within 21 days of PTM-101 placement
  Number of subjects with PTM-101/PTM-101 placement-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Dose Expansion | Within 3 months of PTM-101 placement
  Safety: serious adverse events related to PTM-101 or PTM-101 placement
Dose Expansion | Within 3 months of PTM-101 placement
  Efficacy: volume response rate (VRR) of ≥ 40% reduction in tumor volume
Dose Escalation and Dose Expansion | At 21 days and 3 months post PTM-101 placement
  Overall response rate (ORR) by RECIST 1.1 and WHO
Dose Escalation and Dose Expansion | Within 24 months of PTM-101 placement
  Progression free survival (PFS) per RECIST 1.1
Dose Escalation and Dose Expansion | Within 24 months of PTM-101 placement
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - Northwell Health Zuckerberg Cancer Center, Lake Success, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No